CLINICAL TRIAL: NCT03640065
Title: The Effect of Freeze-Dried Probiotic Sachets Versus Fermented Dairy Product (Yogurt) on Gingival Bleeding on Brushing in Adolescents (12-15) Years Old : A Randomized Clinical Pilot Study
Brief Title: Evaluation of The Effect of Live Probiotic Cultures Present in Fermented Dairy Product (Yogurt) Versus The Effect of Freeze-Dried Probiotic Sachets on Gingival Bleeding of Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Mustafa Samy Ismaiel, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-06-40
Record Dates: First submitted 2018-08-15; First posted 2018-08-21 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Gingival Inflammation
MeSH Terms: conditions — Gingivitis | interventions — Cultured Milk Products; Yogurt

STUDY DESIGN:
Masking Description: only statistician was blind known participants only by codes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- freeze-dried probiotic sachets (Experimental)
  Interventions: Drug: freeze-dried probiotic sachets
- fermented dairy product (yogurt) (Active Comparator)
  Interventions: Dietary Supplement: fermented dairy product ( yogurt)

INTERVENTIONS:
Drug: freeze-dried probiotic sachets — * The participants will be instructed to consume the sachets as follow, each sachet powder is mixed with 10 ml of water in a measuring cup, then swish the mixture in the mouth for one minute before swallowing.
  * This procedure will be repeated once daily for the following 4 weeks.
  * 4 weeks supply will be given to the participants.
  Arms: freeze-dried probiotic sachets
Dietary Supplement: fermented dairy product ( yogurt) — * The participants will be instructed to consume the yogurt once daily regularly for the following 4 weeks.
  * 4 weeks supply will be given to the participants with instruction to store the yogurt in refrigerator at home
  Arms: fermented dairy product (yogurt)

SUMMARY:
To evaluate the effect of probiotics supplied in two different forms (dairy products containing probiotics as yogurt and freeze-dried synthetic probiotics sachets) on improving gingival condition and caries potentiality of dental plaque in adolescents

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 12-15 years old
2. Children complaining from gingival problems
3. Medically free children
4. Children not registered in other clinical researches

Exclusion Criteria:

1. Children with systemic diseases, mental disorders, chronic debilitating diseases.
2. Children using antibiotic treatment during the study
3. Children with orthodontic treatment
4. Children using antimicrobial mouthwash
5. Children taking any probiotic supplemental therapy

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2019-10-20 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Gingival bleeding On Brushing | base line and after 4 weeks
  Patient questioning and answering with yes or no on a questionnaire

SECONDARY OUTCOMES:
Change in Dental plaque pH | base line and after 4 weeks
  Pooled plaque sample (pH meter) on scale (1-14)

CONTACTS AND LOCATIONS:
Locations (1):
- Mai M Ismaiel, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided